CLINICAL TRIAL: NCT01235884
Title: Prevention of the Minor Digestive Disorders by Lactobacillus Reuteri Supplementation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Flavia Indrio, Senior Consultant Neonatologist Pediatric Gastroenterologist, University of Bari
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FI-RF-01/10
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Minor Digestive Disorders
Keywords: gaseous colic, regurgitation and of constipation
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactobacillus reuteri (Active Comparator): Dietary Supplement
  Interventions: Dietary Supplement: Lactobacillus reuteri
- Placebo (Placebo Comparator): Dietary Supplement
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri — 1000000000 CFU per day (5 drops) for 28 days
  Arms: Lactobacillus reuteri
Dietary Supplement: Placebo — 5 drops daily for 28 days
  Arms: Placebo

SUMMARY:
Aim of the study. To evaluate if L. reuteri DSM 17938 supplementation since the first days of life can reduce the onset of gaseous colic in neonates and the onset of minor digestive disorders such as regurgitation and constipation.

Study Design. Double blind, randomized, controlled, multicenter study. 492 neonates of 37-42 gestational age, breast or formula fed, will receive L. reuteri 5 drops (1x108 CFU) daily or placebo for 28 days.

After the inclusion, at baseline will be performed :

* Paediatric visit
* antropometric valutation
* number of the daily crying minutes, number of regurgitation and number of daily evacuation

The patients will receive the probiotics/placebo every days for 28 days and the 29th will be repeated the following analyses:

* Paediatric visit
* antropometric valutation
* number of daily crying minutes
* numbers of regurgitation
* numbers of evacuations

Primary outcome :

To define if Lactobacillus reuteri supplementation can reduce the onset of gaseous colic, regurgitation and of constipation.

Inclusion criteria

* neonates of 37-42 week gestational age and appropriate birth weight
* Recruitment age: until 7 days of life
* Informed consent signed

Exclusion criteria

* Presence of other gastrointestinal diseases.
* Use of FANS, aspirin or other drugs
* Use of antibiotics and/or PPIs e/o anti-H2
* Participation to other clinical trials

ELIGIBILITY:
Inclusion Criteria:

* neonates of 37-42 week gestational age and appropriate birth weight
* Recruitment age: until 7 days of life
* Informed consent signed

Exclusion Criteria:

* Presence of other gastrointestinal diseases.
* Use of FANS, aspirin or other drugs
* Use of antibiotics and/or PPIs e/o anti-H2
* Participation to other clinical trials

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 492 (Actual)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Reduction of the onset of gaseous colic, regurgitation and of constipation. | one year
  After the inclusion, at baseline will be performed :
  * Paediatric visit
  * antropometric valutation
  * number of the daily crying minutes, number of regurgitation and number of daily evacuation
  The patients will receive the probiotics/placebo every days for 28 days and the 29th will be repeated the following analyses:
  * Paediatric visit
  * antropometric valutation
  * number of daily crying minutes
  * numbers of regurgitation
  * numbers of evacuations

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Indrio, MD, Principal Investigator — University of Bari
Locations (8):
- Italy (8):
  - University of Bari, Bari, BA
  - Ospedale Sant'Orsola Malpighi, Bologna, BO
  - Arcispedale S. Anna, Ferrara, FE
  - Ospedale Civile, Crotone, KR
  - Ospedale di Sesto S. Giovanni, Milan, MI
  - Ospedale "SS. Annunziata", Taranto, TA
  - Ospedale "Frà Castoro", San Bonifacio, VR
  - Policlinico "S. Matteo", Pavia

REFERENCES:
- [Derived] Indrio F, Di Mauro A, Riezzo G, Civardi E, Intini C, Corvaglia L, Ballardini E, Bisceglia M, Cinquetti M, Brazzoduro E, Del Vecchio A, Tafuri S, Francavilla R. Prophylactic use of a probiotic in the prevention of colic, regurgitation, and functional constipation: a randomized clinical trial. JAMA Pediatr. 2014 Mar;168(3):228-33. doi: 10.1001/jamapediatrics.2013.4367. PMID 24424513